CLINICAL TRIAL: NCT01325571
Title: A Randomized, Double-blinded, Placebo-controlled, and Multi-centered Clinical Trial Evaluating the Efficacy and Safety of Tacrolimus Capsule in Myasthenia Gravis That Was Insufficiently Treated by Glucocorticoid Therapy
Brief Title: A Study to Compare the Efficacy and Safety of Tacrolimus Capsules in Patient With Myasthenia Gravis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma China, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: F506-CL-0611
Record Dates: First submitted 2011-03-16; First posted 2011-03-30 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-03

CONDITIONS: Myasthenia Gravis
Keywords: prograf; immunosuppressant
MeSH Terms: conditions — Myasthenia Gravis | interventions — Tacrolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- tacrolimus group (Experimental)
  Interventions: Drug: Tacrolimus capsule
- placebo group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tacrolimus capsule — oral
  Other Names: Prograf; FK506
  Arms: tacrolimus group
Drug: Placebo — oral
  Arms: placebo group

SUMMARY:
To evaluate the efficacy and safety of tacrolimus capsules in patients with myasthenia gravis who are inadequately treated by glucocorticoid.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed as myasthenia gravis (MG) by clinical diagnosis
* QMG scores ≥7 at the time of enrollment
* basic treatment drugs are mainly glucocorticoids, and the efficacy of glucocorticoid therapy was not sufficient

Exclusion Criteria:

* receiving blood purification therapy or immunoglobulin therapy within 8 weeks before the study
* QMG swallowing function score ≥ 2 points or QMG vital capacity = 3
* abnormal hepatic functions
* uncontrolled diabetes patients
* hyperkalemia patients
* immuno-inhibitors are forbidden due to malignancy, history of malignancy or history of HIV infection
* patients who are allergic to Tacrolimus or macrolide antibiotics
* receiving other immuno-inhibitors within 12 weeks

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2011-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in quantitative myasthenia gravis (QMG) score for disease severity | Baseline and at 24 weeks
Change from baseline in QMG score for disease severity | Baseline and at 4 weeks
Change from baseline in QMG score for disease severity | Baseline and at 8 weeks
Change from baseline in QMG score for disease severity | Baseline and at 12 weeks
Change from baseline in QMG score for disease severity | Baseline and at 16 weeks
Change from baseline in QMG score for disease severity | Baseline and at 20 weeks

SECONDARY OUTCOMES:
Changes in Osserman classification | Baseline and at 4 weeks, 8 weeks, 12 weeks, 16 weeks, 20 weeks and 24 weeks
Changes in myasthenia gravis activity of daily living scale | Baseline and at 4 weeks, 8 weeks, 12 weeks, 16 weeks, 20 weeks and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (9):
- China (9):
  - Beijing
  - Guangdong
  - Jiangsu
  - Jilin
  - Shandong
  - Shanghai
  - Sichuan
  - Wuhan
  - Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhou L, Liu W, Li W, Li H, Zhang X, Shang H, Zhang X, Bu B, Deng H, Fang Q, Li J, Zhang H, Song Z, Ou C, Yan C, Liu T, Zhou H, Bao J, Lu J, Shi H, Zhao C. Tacrolimus in the treatment of myasthenia gravis in patients with an inadequate response to glucocorticoid therapy: randomized, double-blind, placebo-controlled study conducted in China. Ther Adv Neurol Disord. 2017 Sep;10(9):315-325. doi: 10.1177/1756285617721092. Epub 2017 Jul 26. PMID 28861121
- See also: Link to results on Astellas Clinical Study Results Web site — https://www.astellasclinicalstudyresults.com/hcp/study.aspx?ID=F506-CL-0611